CLINICAL TRIAL: NCT05112003
Title: Translingual Neurostimulation for the Virtual Treatment of Post-Traumatic Stress Disorder: A Feasibility Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthTech Connex Inc. (Industry)
Collaborators: Centre for Neurology Studies (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTC_PTSD_001
Record Dates: First submitted 2021-10-15; First posted 2021-11-08 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TLNS (Experimental): Translingual neurostimulation will be paired with breathing and awareness training prior to CPT sessions
  Interventions: Device: Translingual neurostimulation
- Control (No Intervention): No TLNS

INTERVENTIONS:
Device: Translingual neurostimulation — The device will be placed into and held in the participant's mouth for 20 minutes while the participant undergoes breathing and awareness training
  Arms: TLNS

SUMMARY:
A growing body of evidence suggests that translingual neurostimulation (TLNS) plays a role in modulating neuroplastic changes in the brain, which has far-reaching implications for its ability to facilitate other therapeutic interventions such as cognitive processing therapy (CPT) for post-traumatic stress disorder (PTSD). The present study aims to assess the feasibility of combining TLNS with CPT in individuals with PTSD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 19 years of age or older
2. A score of 33 or more on the Posttraumatic Stress Disorder Checklist (PCL-5)
3. PTSD symptom duration of ≥ 12 months
4. Stable dose of any medications for the last three months, with no changes anticipated for the duration of the study
5. Adequate support at home (e.g., family member or caregiver) to ensure assistance in seeking access to help if needed
6. Able to understand the informed consent form, study procedures and willing to participate in study
7. Currently has a primary care provider

Exclusion Criteria:

1. History of substance dependence or abuse (within the last 3 months)
2. Unstable psychosocial settings (homelessness, lack of support at home)
3. Moderate to high risk of suicidal ideation or behaviour as measured by the Columbia Suicide Severity Rating Scale (C-SSRS)
4. Current diagnosis of severe anxiety (or score of ≥15 on the GAD-7), severe depression (or score of ≥20 on the PHQ-9), schizophrenia or bipolar disorder
5. Use of medications for PTSD within the last 6 weeks
6. History of other major neurological disorder (brain cancer, dementia, multiple sclerosis, stroke)
7. Detection of mild cognitive impairment (mini-ACE score of ≤ 25)
8. Diagnosed epilepsy or history of seizures
9. Not proficient in English
10. Recent (within last 2 years) acquired brain injury
11. Exposed to an investigational drug or device 30 days prior to starting the study, or concurrent use of an investigational drug or device while enrolled in the study
12. If female and of child-bearing potential: pregnant, suspected or planning to become pregnant or breast-feeding
13. Contraindicated for the NeuroCatchTM Platform, including:

    13.1. Requires the use of hearing aids or a cochlear implant 13.2. Diagnosed with tinnitus that is currently active 13.3. Has temporary damage to earing (e.g. punctured ear drum) 13.4. Unable to detect a 740Hz tone played at 85dB in both ears. 13.5. Implanted pacemaker or implanted electrical stimulators 13.6. Metal or plastic implants in the skull, excluding dental/facial implants 13.7. Unhealthy scalp (apparent open wounds and/or bruised or weakened skin) 13.8. Previous exposure to the NeuroCatch™ Platform audio sequences in the last 3 months
14. Contraindicated for PoNSTM use, including:

14.1. Current disease or sensitivity of the oral cavity 14.2. History of oral cancer 14.3. Oral surgery within three months of screening 14.4. Oral cavity piercings that could interfere with PoNSTM use 14.5. Sensitivity to Nickel, Copper, or Gold 14.6. Currently enrolled in a PoNSTM treatment program or use of the PoNSTM device in the last 5 weeks 14.7. History of penetrating brain injuries 14.8. History of neurodegenerative diseases 14.9. Chronic infectious disease 14.10. Unmanaged hypertension 14.11. Diabetes 14.12. History of seizures

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Proportion of participants screened who are eligible | Baseline to week 6
  Reach (RE-AIM framework)
Clinician-rated symptom severity as measured by CAPS | Change from baseline to week 6
  Effectiveness (RE-AIM framework)
Participant rated symptom severity as measured by the PCL-5 | Change from baseline to week 6
  Effectiveness (RE-AIM framework)
Proportion of therapy visits completed | Baseline to Week 6
  Adoption (RE-AIM framework)
Ease of protocol administration | Baseline to week 6
  Adoption (RE-AIM framework); 5-point Likert scale for participants and therapists
Qualitative report of barriers and facilitators | Baseline to week 6
  Implementation (RE-AIM framework)

SECONDARY OUTCOMES:
Electroencephalography (EEG) | Change from baseline to week 6
  Using the NeuroCatchTM Platform - EEG amplitudes
Electroencephalography (EEG) | Change from baseline to week 6
  Using the NeuroCatchTM Platform - EEG latencies
Generalized Anxiety Disorder 7-item (GAD-7) | Change from baseline to week 6
  Anxiety symptom severity self-report measure
Patient Health Questionnaire (PHQ-9) | Change from baseline to week 6
  Depression symptom severity self-report measure
Brief Inventory of Psychosocial Functioning (B-IPF) | Change from baseline to week 6
  PTSD-related functional impairment in the prior 30 days
Meaning in Life Questionnaire (MLQ) | Change from baseline to week 6
  Assesses two dimensions of meaning in life using 10 items rated on a seven-point scale
Time from inciting event | Baseline
  Time since traumatic event (years)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Neurology Studies, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study sign-up page — https://centreforneurologystudies.com/neurostimulation-therapy-for-post-traumatic-stress-disorder/